CLINICAL TRIAL: NCT02955498
Title: A Randomized, Open-label, Single-Dose, 2-Treatment, 2-Way, 2-Period Crossover Study to Assess the Safety and the Pharmacokinetic Characteristics of Lodivikar Tab. 5/40 mg in Healthy Adult Male Subjects
Brief Title: Clinical Trial to Assess the Pharmacokinetic Characteristics of Lodivikar Tab. 5/40 mg in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HL-LVK-101
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-T (Experimental): First period: administration of reference drug, Second period: administration of test drug
  Interventions: Drug: Sevikar tab. 10/40mg; Drug: Lodivikar tab. 5/40mg
- T-R (Experimental): First period: administration of test drug, Second period: administration of reference drug
  Interventions: Drug: Sevikar tab. 10/40mg; Drug: Lodivikar tab. 5/40mg

INTERVENTIONS:
Drug: Sevikar tab. 10/40mg — Reference drug: Sevikar tab. 10/40mg, 1T, single oral administration in the fasted state
Drug: Lodivikar tab. 5/40mg — Test drug: Lodivikar tab 5/40mg, 1T, single oral administration in the fasted state

SUMMARY:
The purpose of this study is to assess the pharmacokinetic characteristics of olmesartan and S-amlodipine after single oral administration of Sevikar tab. 10/40mg, a combination formulation of olmesartan and amlodipine as reference drug and Lodivikar tab. 5/40mg, a combination formulation of olmesartan and S-amlodipine as test drug in healthy male adults. Additionally the safety and tolerability of two drugs will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male in the age of 20-45
* Body weight ≥ 55kg, IBW ± 20%
* Subject who sign on an informed consent form willingly

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with known for hypersensitivity reaction to S-amlodipine, amlodipine and olmesartan and dihydropyridine derivatives
* Clinically significant hypotension (SBP≤100mmHg, DBP≤60mmHg) or hypertension(SBP≥150mmHg, DBP≥95mmHg) when screening period
* Subject with known for history of disease or gastric surgery which affect on the absorption,
* Subject with any of the following conditions in laboratory test

  * AST or ALT > UNL (upper normal limit) x 1.5
  * Total bilirubin > UNL x 1.5
  * Renal failure with CLcr < 50mL/min calculated on Cockcroft-Gault [Cockcroft-Gault GFR = (140-age) * (Wt in kg) / (72 *Cr)]
  * Serum potassium < 3.5 mEq/L or > 5.5 mEq/L
* Continued excessive use of caffeine (caffeine >five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker(cigarette >10 cigarettes per day)
* Participation in any clinical investigation within 60days prior to study medication dosing
* Subject with whole blood donation within 60days, component blood donation within 30days prior to study medication dosing
* Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28days prior to study medication dosing
* Use of any prescription medication including oriental medication within 14 days prior to study medication dosing or over-the-counter medication within 7 days prior to study medication dosing
* Subject with mental illness or drug addiction
* Subject taking foods which affect on the absorption, distribution, metabolism or excretion of drug within 7days prior to study medication dosing
* Subject with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144hr(19 points)
Peak Plasma Concentration (Cmax) | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144hr(19 points)

SECONDARY OUTCOMES:
Number of participants with adverse events | From study medication dosing day to follow-up period for maximum 7 days from the second period discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Metrohospital, Anyang, Kyung Gi, South Korea